CLINICAL TRIAL: NCT05569876
Title: Vocal Biomarkers for the Detection and Prevention of Hypoglycemia (HypoVoice)
Brief Title: The HypoVoice Study
Acronym: HypoVoice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Idiap Research Institute (Unknown); CSEM Centre Suisse d'Electronique et de Microtechnique SA (Unknown); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HypoVoice
Record Dates: First submitted 2022-09-22; First posted 2022-10-06 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus; Hypoglycemia
Keywords: Hypoglycemia; Voice; Speech; Detection; Artificial intelligence (AI)
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Speech

STUDY DESIGN:
Masking Description: Participants are aware that hypoglycemia will be induced during the study but they are blinded to their blood glucose levels throughout the hypoglycemia procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled hypoglycemic state (Other)
  Interventions: Other: Controlled hypoglycemic state

INTERVENTIONS:
Other: Controlled hypoglycemic state — Voice sampling is performed in different glycemic states (euglycemia and hypoglycemia).

SUMMARY:
The HypoVoice study aims at identifying potential vocal biomarkers associated with hypoglycemia to pave the way towards a voice-based hypoglycemia detection approach.

DETAILED DESCRIPTION:
While hypoglycemia has been widely studied in medical research, studies assessing vocal changes associated with this state are limited. This study aims at collecting a data set labelled with the gold standard (blood glucose) to provide a solid basis for the identification of vocal biomarkers using machine learning. Additionally, physiological data are collected using wearable sensors to assess whether additional integration of vital signs (e.g. heart rate) enhances the performance of hypoglycemia detection.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Type 1 Diabetes mellitus as defined by WHO for at least 6 months
* Aged 18 - 60 years
* HbA1c ≤9.0 %
* Functional insulin treatment with good knowledge of insulin self-management
* Native language German or Swiss German
* Use of continuous glucose monitoring (CGM) or flash glucose monitoring (FGM)

Exclusion Criteria:

* Incapacity to give informed consent
* Contraindications to insulin aspart (NovoRapid®)
* Total daily insulin dose >2 IU/kg/day
* Pregnancy, breast-feeding or lack of safe contraception
* Active heart, lung, liver, gastrointestinal, renal or psychiatric disease
* Pacemaker or implantable cardioverter defibrillator (ICD)
* Epilepsy or history of seizure
* Chronic neurological or ear-nose-and-throat (ENT) disease influencing voice or history of voice disorder
* Illiteracy or dyslexia
* Active smoking
* Active drug or alcohol abuse
* Medication known to interfere with voice or to induce listlessness (e.g. opioids, benzodiazepines, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the HypoVoice approach to detect hypoglycemia based on voice data quantified as area under the receiver operating characteristic curve (AUROC) | 4 hours
  Voice data will be collected in eu- and hypoglycemia

SECONDARY OUTCOMES:
Diagnostic accuracy of the HypoVoice approach to detect hypoglycemia based on voice and physiological data quantified as area under the receiver operating characteristic curve (AUROC) | 4 hours
  Voice and physiological data will be collected in eu- and hypoglycemia
Voice parameters indicative of hypoglycemia | 4 hours
  Explainable AI methods will be used to identify voice parameters indicative of hypoglycemia
Physiological parameters indicative of hypoglycemia | 4 hours
  Explainable AI methods will be used to identify physiological parameters indicative of hypoglycemia

OTHER OUTCOMES:
Change in hypoglycemic symptoms across the glycemic trajectory | 4 hours
  Hypoglycemic symptoms will be assessed using the Edinburgh Hypoglycemia Scale (higher score means more symptoms).
Change in cognitive performance across the glycemic trajectory. | 4 hours
  Cognitive performance will be assessed using the Digit Symbol Substitution Test (higher score means better cognitive performance).
Change in cognitive performance across the glycemic trajectory. | 4 hours
  Cognitive performance will be assessed using the Trail Making B Test (more time needed to complete the tests means worse cognitive performance).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Prof. MD, Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Bern, Switzerland